CLINICAL TRIAL: NCT02855866
Title: Interest of Cryotherapy or Cortisone Aerosol Therapy in Early Post-operative Swallowing Disorders Following Total Thyroidectomy
Acronym: DEGLUTHYR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: OSMAK POUSSIER 2013
Record Dates: First submitted 2016-07-28; First posted 2016-08-04 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Thyroidectomy; Post-operative Swallowing Disorders
MeSH Terms: interventions — Thyroidectomy; Cryotherapy; dexamethasone acetate; Acetaminophen

ARMS (3):
- cryotherapy (Experimental)
  Interventions: Procedure: thyroidectomy; Other: cryotherapy; Drug: Dexamethasone acetate; Drug: paracetamol
- Cortisone aerosol (Active Comparator)
  Interventions: Procedure: thyroidectomy; Drug: cortisone aerosol; Drug: Dexamethasone acetate; Drug: paracetamol
- Management (Placebo Comparator)
  Interventions: Procedure: thyroidectomy; Drug: Dexamethasone acetate; Drug: paracetamol

INTERVENTIONS:
Procedure: thyroidectomy
Other: cryotherapy
  Arms: cryotherapy
Drug: cortisone aerosol
  Arms: Cortisone aerosol
Drug: Dexamethasone acetate
Drug: paracetamol

SUMMARY:
The scientific interest of this study is to improve post-operative comfort in patients after thyroid surgery using simple, inexpensive techniques. The investigator expects that local applications of ice or cortisone aerosols will reduce swallowing discomfort and control post-operative pain (POP). The investigator hopes that local cryotherapy will decrease post-operative oedema (vasoconstriction) and the volume of liquid drained (action on the serous fluid at the site of the thyroidectomy).

ELIGIBILITY:
Inclusion Criteria:

* Patients about to undergo total thyroidectomy by cervicotomy
* Single surgeon: Dr Osmak-Tizon Liliana
* Patients who have provided written consent to take part in the research
* Hospitalized in the endocrine surgery unit
* Whose mental and physical state allows them to participate in the quantification of a symptom using a Visual Analogue Scale(VAS)

Exclusion Criteria:

* Patients under 18 or adults under guardianship
* Patients about to undergo unilateral thyroid surgery (thyroid lobectomy)
* Patient who have had parathyroid surgery
* History of cervicotomy
* Intolerance to, contra-indication for or allergy to any of the treatments tested.
* Pregnant or breast-feeding women
* Patients without national health insurance cover

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2013-09-03 (Actual); Primary Completion 2015-02-20 (Actual); Study Completion 2015-02-20 (Actual)

PRIMARY OUTCOMES:
Swallowing Impairment Score (SIS). | Evolution of the SIS from baseline (inclusion), to the end of the surgery and every day thereafter until discharge of the patient(up to 3 months)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France